CLINICAL TRIAL: NCT02821663
Title: Rehabilitation in Patients Suffering From Systemic Sclerosis by Vocal Intervention: A Pilot Study
Brief Title: Vocal Intervention in Systemic Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Michael Mickel, MD, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SSc-1-MM
Record Dates: First submitted 2016-06-24; First posted 2016-07-01 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Systemic Sclerosis
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vocal intervention (Experimental): Vocal intervention
  Interventions: Behavioral: vocal intervention

INTERVENTIONS:
Behavioral: vocal intervention — 10 x 60 min. sessions of vocal intervention

SUMMARY:
Systemic sclerosis is a systemic connective tissue disease with physical and mental disturbances. Based on a pilot study the feasibility and effectiveness of a novel, self-developed concept of vocal intervention in Systemic Sclerosis under vocal pedagogical guidance and music therapy is assessed.

DETAILED DESCRIPTION:
This concept aims at functional improvement of respiration and mouth-opening, enhancement of Quality of Life, and reduction of stress carried out by a music therapist and singer with pedagogical formation.

ELIGIBILITY:
Inclusion Criteria:

* positive criteria for Systemic Sclerosis according to the American College of Rheumatology/European League Against Rheumatism

Exclusion Criteria:

* affection of the vocal apparatus
* dyspnea at rest
* oxygen prescription

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2014-11; Primary Completion 2017-10 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
MOS 36-Item Short Form Health Survey | up to 4 weeks
  The SF-36 - a patient-reported survey of patient health - consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight.

SECONDARY OUTCOMES:
Mouth open; in millimeter | up to 4 weeks
  incisor to incisor; corner of mouth to corner of mouth; measurement by tape
6-minutes walk test | up to 4 weeks
  The 6-minute walk test assess changes in functional exercise capacity with the primary outcome reported being the distance walked during the test.
Secretory immunoglobulin A; mg/l | up to 4 weeks
  Immunoglobulin A is an antibody that plays a role in immune function in the mucous membranes. Indicates changes in immune status. Collected by a swab placed in the mouth.
Saliva cortisol; ng/ml | up to 4 weeks
  Cortisol is a steroid hormone indicating changes in stress status. Collected by a swab placed in the mouth.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Mickel, MD, Principal Investigator — Deptartment of Physical Medicine and Rehabilitation, MUW
Locations (1):
- Department of Physical Medicine and Rehabilitation, Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided